CLINICAL TRIAL: NCT00998114
Title: Early Detection of Diastolic Dysfunction and the Role of Lifestyle Measures in Its Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Anand Chockalingam, Prof Assoc, Medicine-Cardiology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1115737
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Diastolic Dysfunction
Keywords: Early Cardiac Diastolic Dysfunction; Aerobic Exercise; Weight Reduction
MeSH Terms: conditions — Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise and diastolic dysfunction (Experimental): Aerobic exercise for 30-45 minutes five times a week for six months
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Aerobic exercise for 30-45 minutes five times a week for six months
  Other Names: Diastolic Dysfunction

SUMMARY:
The project aims to investigate the effect of a regular exercise for 6 months on diastolic parameters in patients who present with shortness of breath and who have evidence of early diastolic dysfunction on echocardiography. Patients will be enrolled from the VA General Medicine and Cardiology Clinics, and will be screened for diastolic dysfunction. Once enrolled, they will be on an exercise regimen that involves aerobic exercise for 30-45 minutes five times a week at home. The participants will have an initial supervised exercise session with the VA Cardiac Rehabilitation team, and will have either every other week or monthly supervised sessions at the VA Cardiac Rehabilitation Center to monitor their progress. Clinical, biometric, laboratory and echocardiographic parameters will be obtained before and after the 6 month period.

DETAILED DESCRIPTION:
Introduction:

Diastolic dysfunction (DD) accounts for >50% of all heart failure (DHF) hospitalizations and this number is increasing with age, obesity and diabetes.

There are no proven treatments for DHF apart from blood pressure control.

Aim:

If diagnosed early, is this reversible with lifestyle changes; namely, aerobic exercise and weight reduction?

Methods:

We will screen veterans presenting to the medicine, cardiology and pulmonary services with dyspnea. We will perform echocardiography with Doppler which non-invasively measures cardiac filling and diastolic dysfunction. Treadmill exercise echo will be performed to quantify DD.

Bruce treadmill protocol description/ procedure: Exercise is performed on a treadmill. The test starts at 2.74 km/hr (1.7 mph) and at a gradient (or incline) of 10%. At three minute intervals the incline of the treadmill increases by 2%, and the speed increases as shown in the table below.

Stage Speed (mph) Gradient:

1. 1.7 10
2. 2.5 12
3. 3.4 14
4. 4.2 16
5. 5.0 18
6. 5.5 20
7. 6.0 22
8. 6.5 24
9. 7.0 26
10. 7.5 28

Subject exercise study:

For physical exercise to have a beneficial effect on cardiac function, we suggest the following:

* Type of Exercise
* Walking - outdoors or treadmill
* Running or jogging
* Cycling - outdoors or stationary

Duration of Exercise:

Initial 2-3 minute gradual warm-up period. Roughly 30 minutes of continuous exercise 5 times a week.

Finally a few minutes of gradual cool-down before terminating exercise.

Intensity of Exercise:

Target exercise at a "moderately significant exertion".

We will demonstrate what is adequate in the beginning and periodically throughout the 6 months of the study.

"Maximum age predicted heart rate (MPHR)" is calculated as 220 minus subject's age. Then we would like to sustain roughly about 70 to 85% of MPHR for 25-30 minutes.

"Successful" Exerciser: Subjects who are able to adhere to the required intensity and duration of exercise for the majority (about 75% or more) of the time; averaging 150 minutes/ week on self reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspnea/shortness of breath
* Age 40-65 years of age
* Sedentary lifestyle (<150 minutes of exercise/week)
* Echocardiographic evidence of early diastolic dysfunction: mitral E/A <0.9, OR resting E/E' between 8-15 cm/s, OR post-exercise E/E' >13 cm/s.

Exclusion criteria:

* Age <40 years or >65 years
* Coronary Artery Disease by angiography or evidence of ischemia on a stress test
* Systolic Dysfunction (LV Ejection fraction <50%)
* Congestive Heart Failure Functional Class III or IV
* Moderate to severe COPD (FEV <80% predicted)
* Moderate to severe valvular heart disease, except tricuspid regurgitation
* Inability to get heart rate >/= 85% of maximum predicted heart rate
* Uncontrolled hypertension (systolic BP>140mmHg, diastolic BP>90mmHg) despite medical therapy
* On echocardiogram, RV systolic pressure >60mmHg that suggests severe pulmonary hypertension
* On echocardiogram, left atrial size> 6.5 cm or left atrial volume > 35 ml/BSA

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Exercise echo Doppler will be done at baseline and after completion of 6 months of an exercise program | Beginning of study participation and after 6 months of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Anand Chockalingam, MD, Principal Investigator — University of Missouri/Harry S Truman VA Hospital
Locations (1):
- Harry S Truman Veterans Administration Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No